CLINICAL TRIAL: NCT05123014
Title: Lenticule Implantation and Autologous Serum New Approach in Treatment of Adenoviral Keratitis Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EyeHPristina 1
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-02

CONDITIONS: Adenoviral Keratoconjunctivitis

STUDY DESIGN:
Intervention Model Description: LENTICULE IMPLANTATION AND AUTOLOGOUS SERUM NEW APPROACH IN TREATMENT OF ADENOVIRAL KERATITIS DISEASE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ReLex Smile surgery (Other): Fresh Corneal Lenticule Implantation using Relex-Smile Surgery We used all preoperative procedures atlas, optic tomography and especially electron microscope. Approximately we planned how much microns we remove and insert with the purpose to remove more dead keratocytes which increase biomechanical instability of corneal metabolism (abnormal increase collagenase activity, decrease proteinase inhibitors, excessive premature keratocyte apoptosis, increase cytokine binding). Fresh Corneal Lenticule and autologous serum contains live stem cells that produce keratocytes, collagen fibers, extracellular matrix which contribute to the regeneration of the cornea, and all this results at increasing of corneal transparency and visual acuity in patients with adenoviral keratitis.
  Interventions: Other: relex smile

INTERVENTIONS:
Other: relex smile — In OCT, firstly, the thickness of the adenoviral subepithelial infiltration in the cornea is calculated in microns, and extraction is performed accordingly with Small Incision Lenticule Extraction( SMILE )and fresh lenticule implanted stromal in the same volume.

SUMMARY:
Adenoviral keratitis(caused by adenovirus) is one of the most frequently diagnosed eye diseases. Most of these infections have symptoms like (Ocular itchiness and irritation, chemosis (conjunctival edema),photophobia, epiphora, foreign body sensation, epithelial keratitis etc.Adenoviral subepithelial infiltration is one of the most difficult complication to treat. Our purpose is to evaluate corneal transparency, recurrence, and visual acuity in patients with adenoviral subepithelial infiltration by first removing the infiltrative stroma with a smile and implanting the same volume of fresh lenticule in the prepared stromal pocket.

DETAILED DESCRIPTION:
Our treatment of adenoviral keratitis using lenticule implantation and autologus serum it has been applied to patients who have received medical treatment(Antiviral medications, topical corticosteroids ,compresses, artificial tears, and topical cycloplegic) for a long time but have not been successful.

In OCT, firstly, the thickness of the adenoviral subepithelial infiltration in the cornea is calculated in microns, and extraction is performed accordingly with Small Incision Lenticule Extraction( SMILE )and fresh lenticule implanted stromal in the same volume. AS-OCT was evaluated using corneal topography and glass-corrected best visual acuity (BSCVA) measurements and electron microscopy. Postoperative complications were recorded during the follow-up period.

The patients were followed for one year. No complications were observed in the patients. After the operation, there was an increase in satisfaction and vision. They returned to their daily lives very quickly.

Postoperatively, uncorrected vision increased to 6 lines in 12 eyes, seven lines in 11 eyes, and eight lines in 3 eyes.

ELIGIBILITY:
Inclusion Criteria:

* low transparency of cornea
* low visual acuity
* recurrence keratitis

Exclusion Criteria:

* active anterior segment pathology
* previous corneal or anterior segment surgery
* any infection

Ages: 24 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Increasing corneal transparency | 12 months
  Implanting lenticule with stromal stem cells ,live keratocytes and putting autologous serum to stabilize biomechanical stability of cornea.

SECONDARY OUTCOMES:
Increase of visual acuity | 12 months
  Upon implanting fresh corneal lenticule according to clarity of cornea, uncorrected vision increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No